CLINICAL TRIAL: NCT02734394
Title: UW WELL-FIT Exercise Program for Cancer Patients
Acronym: WELL-FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Julia Fraser, Research and Operations Manager, University of Waterloo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ORE18987-A
Record Dates: First submitted 2016-02-09; First posted 2016-04-12 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: exercise; body composition; metabolism; nutrition
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular and strength training exercise (Experimental): 24 sessions (~12 weeks) exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Cardiovascular and resistance exercise training

SUMMARY:
The purpose of this project is to help to manage the many cancer treatment side effects through cardiovascular and resistance exercise, and education with the goal of using program outcomes to contribute to current research.

DETAILED DESCRIPTION:
This study is a single group pre-test post-test design.There are 4 optional measures that will be presented to participants from which they can choose to participate or not. These are presented with check boxes in the consent form. After completion of the University of Waterloo (UW) WELL-FIT program, participants will be given an option to continue with an exercise program; they will be offered the Graduate Program. Following consent of Graduate Program, repeated measures would be taken annually. At the time of consent, they will have the option to have their data used in research. At any point in their involvement of the exercise based programs, they can indicate "they no longer want to participate in the program or the data collection". Their medical care or participation in the UW WELL-FIT program will not be affected.

Procedures

1. UW WELL-FIT advertisement for Grand River Regional Cancer Centre
2. UW WELL-FIT brochure
3. Referral Form
4. Participants initial consultation and assessment
5. Obtain consent for UW WELL-FIT
6. Obtain Participant Information
7. Completion of FACIT-F survey
8. Metabolism & Body Composition - Information sheet for optional measures
9. Physical Activity Survey- Godin Questionnaire
10. Provide 3-Day food diary and Nutritional Assessment
11. Fitness assessment, exercise programming and data entry:

    1. Submaximal cardiovascular cycle ergometer or treadmill graded exercise test
    2. Muscular strength using force transducer
    3. Body composition:

       * Height, weight and waist girth
       * Bioelectrical Impedance Analysis (BIA)
       * Dual Energy X-ray Absorption (Optional)
    4. Range of motion using a goniometer
    5. Blood sampling (Optional)
    6. Design Individualized exercise program
12. UW WELL-FIT - Commencement of participant in 12 week exercise program (2 x 60 minute classes)
13. Post assessment (repeated pre-test assessments)
14. Pre and post data are entered into database
15. Summary and Feedback Report
16. Graduate Program: participant selects to attend UW WELL-FIT Graduate Program
17. Participants have annual reassessments in the Graduate Program

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with cancer and will currently be receiving some form of treatment (chemotherapy, radiation therapy or hormonal therapy)

Exclusion Criteria:

* Physical / health factors that prohibit exercise or lack of medical clearance from physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximal Exercise Test | 24 sessions (12 weeks)
  Pre and post maximum workload using an electronic cycle ergometer in Watts
Upper and Lower Limb Strength | 24 sessions (12 weeks)
  pre and post strength in upper and lower limb muscles using a linear differential variable transducer (LVDT) measured in Newton.meters
Body Mass Index | 24 sessions (12 weeks)
  Pre and post body mass index (kg/m2)
Percent Body Fat | 24 sessions (12 weeks)
  Pre and Post percent body fat (units: %)

SECONDARY OUTCOMES:
Glucose | 24 sessions (12 weeks)
  measurement of blood glucose in mM
Lipids | 24 sessions (12 weeks)
  measurement of total cholesterol, low density lipoprotein,high density lipoprotein ( millimole per liter (mM/L)

CONTACTS AND LOCATIONS:
Overall Officials: Caryl Russell, MSc, Principal Investigator — University of Waterloo; Michael Sharratt, PhD, Principal Investigator — University of Waterloo; Marina Mourtzakis, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No